CLINICAL TRIAL: NCT06002672
Title: Analysis of the Potential Health Effects of Saline Eustress in Plant Food
Brief Title: Effects of Saline Eustress in Plant Food (ESEPF)
Acronym: ESEPF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Sara Baldassano, Professor, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Plant_Food_2021
Record Dates: First submitted 2023-07-14; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Healthy Diet
MeSH Terms: interventions — Soil; Water

STUDY DESIGN:
Intervention Model Description: control vs intervention
Who Masked: Participant, Investigator
Masking Description: Two groups that consumed lettuce. No differences in shape, size, colours of lettuce
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): group that consumed control lettuce
  Interventions: Dietary Supplement: Placebo comparator: Control group. To the control group was assigned lettuce without any change in salinity but with the same characteristic of eustress lettuce (soil, water, harvesting time).
- Intervention (Active Comparator): group that consumed eustress lettuce
  Interventions: Dietary Supplement: Experimental: Eustress group. To the intervention Eustress group was assigned the eustress lettuce.

INTERVENTIONS:
Dietary Supplement: Placebo comparator: Control group. To the control group was assigned lettuce without any change in salinity but with the same characteristic of eustress lettuce (soil, water, harvesting time). — Lettuce without any eustress was assigned to each participant belonging to the control group which ate 100gr every day for 12 day
  Other Names: control lettuce
  Arms: Control
Dietary Supplement: Experimental: Eustress group. To the intervention Eustress group was assigned the eustress lettuce. — 100gr of eustress lettuce were assigned to each participant belonging to the intervention group which ate 100 grams every day for a total of 12 days
  Other Names: Eustress Intervention group
  Arms: Intervention

SUMMARY:
The aim of the project is to study if supplementation with eustress plant food like lettuce grown in mild salinity condition affects health in a healthy population.

DETAILED DESCRIPTION:
Salinity can affect the levels of bioactive compounds in leafy vegetables. The aim of the project is to verify the impact, if any, of the changing of bioactive compounds in the physiology of the study population. The participants will be randomly assigned to the control group that will eat 100 gr of untreated (control) lettuce and the intervention group that will consume 100gr of eustress lettuce. Blood samples and urine samples will be collected at time zero (start) after 12 days. Each subject will be subjected to two venous blood samples taken at the beginning of the observation and at the end. The samples obtained will be transported in certified containers for the safe transport of biological samples, and, subsequently, processed by the experimenters at the laboratories of the Molecular Biology section of the University of Palermo. Serum and plasma will be obtained from each blood sample. All information thus obtained will be recorded in a database in which each person will be identified with a numerical code, in order to comply with current privacy regulations. Body weight, Barefoot standing height, Body mass index, Body composition will be measured in the different groups of study. Samples will be analyzed and compared for glucose, insulin, albumin, total cholesterol, HDL-cholesterol, LDL-cholesterol, triglycerides, AST, ALT, GGT, ALP, Ferritin, free Iron, transferrin, total proteins, magnesium, calcium, insulin, osteocalcin, calcitonin, parathyroid hormone, c terminal peptide of collagen (CTX), Vitamin D, Phosphate, Potassium.

ELIGIBILITY:
Inclusion Criteria:

* Italian
* age: 18-65 years
* currently injury free
* Body mass index between 18.5 and 28 kg/m2

Exclusion Criteria:

* Use of vitamins and minerals supplements,
* use of medications
* Presence of metabolic or chronic disease
* Pregnancy, breastfeeding condition,
* smokers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
anthropometric measurement | 12 days
  weight in kilograms, height in meters will be aggregated to arrive at one reported value (weight and height will be combined to report BMI in kg/m^2).
Bone metabolism markers | 12 days
  Parathyroid hormone (PTH) (ng/ml), calcitonin (ng/ml) will be assessed at baseline and after 12 days.
Vitamin D | 12 days
  Vitamin D (microgram/L) will be assessed at baseline and after 12 days.
blood markers | 12 days
  Calcium (mg/dL), Phosphate (mg/dL) will be assessed at baseline and after 12 days.
Potassium | 12 days
  Potassium (mmol/L) will be assessed at baseline and after 12 days.
Bone remodelling markers | 12 days
  markers of bone resorption CTX (μg/L) and bone formation osteocalcin (μg/L) will be assessed in serum at baseline and after 12 days.
Iron | 12 days
  iron (μg/dL) will be assessed in serum at baseline and after 12 days.
Ferritin | 12 days
  ferritin (ng/dL) will be assessed in serum at baseline and after 12 days.
transferrin | 12 days
  transferrin (mg/dL) will be assessed in serum at baseline and after 12 days.
% saturation of transferrin | 12 days
  % saturation of transferrin will be will be assessed in serum at baseline and after 12 days.
markers of lipid metabolism | 12 days
  triglycerides , HDL, LDL, cholesterol (in mg/dL) will be measured in serum will be assessed at baseline and after 12 days.
Insulin | 12 days
  insulin (mUI/L) will be measured in serum will be assessed at baseline and after 12 days.
Glucose | 12 days
  Glucose (mg/dL) will be measured in serum will be assessed at baseline and after 12 days.
markers of hepatic metabolism | 12 days
  Aspartate transaminase (AST), Alanine aminotransferase (ALT), Alkaline phosphatase (ALP), Gamma-Glutamyl Transferase (GGT) in U/l will be assessed in serum at baseline and after 12 days.
Total protein (TP) and Albumin | 12 days
  Total protein (TP) and Albumin in g/L will be assessed in serum at baseline and after 12 days.

SECONDARY OUTCOMES:
body composition | 12 days
  lean mass as percent of body weight and fat mass as percent of body weight will be will be assessed at baseline and after 12 days

CONTACTS AND LOCATIONS:
Overall Officials: Sara Baldassano, Principal Investigator — University of Palermo
Locations (1):
- NABbio, STEBICEF department, Palermo, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ferrantelli V, Vasto S, Alongi A, Sabatino L, Baldassano D, Caldarella R, Gagliano R, Di Rosa L, Consentino BB, Vultaggio L, Baldassano S. Boosting plant food polyphenol concentration by saline eustress as supplement strategies for the prevention of metabolic syndrome: an example of randomized interventional trial in the adult population. Front Nutr. 2023 Dec 22;10:1288064. doi: 10.3389/fnut.2023.1288064. eCollection 2023. PMID 38196756